CLINICAL TRIAL: NCT00155558
Title: A Phase I Trial of HDFL48(Weekly 48-Hour Infusion of High-Dose 5-Fluorouracil and Leucovorin) in Recurrent or Metastatic Colorectal Cancers
Brief Title: A Phase I Trial of HDFL48 in Recurrent or Metastatic Colorectal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 159I13
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2000-11

CONDITIONS: Recurrent or Metastatic Colorectal Cancer
Keywords: Colorectal Cancer, Maximum tolerated dose
MeSH Terms: conditions — Recurrence; Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: 5-Fluorouracil, Leucovorin

INTERVENTIONS:
Drug: 5-Fluorouracil, Leucovorin

SUMMARY:
To determine the maximum tolerated dose and dose limiting toxicity of 5-FU and leucovorin with novel 48-hour infusion schedule, and to collect toxicity profile at different dose level of 5-FU/LV 48-hour infusion.

DETAILED DESCRIPTION:
Colorectal cancer is one of the major in Taiwan.It caused 3128 deaths in 1999, and represented the No.3 cancer killer in both male and female population of Taiwan.

Recently, evidence has accumulated that weekly, 24-hour infusion of high-dose 5-FU may improve the response rate and survival time compared with 5-FU bolus regiment. In a randomized multicenter trial of metastatic colorectal cancer, Kohne et al reported an overall response rate of 44%and a median survival time of 16 months using a weekly-times-six schedule of infusional 5-FU (2600mg/m2 24-hours infusion). In another randomized study for advanced colorectal cancer, de Gramont et al reported a significantly better outcome in patients treated by a similar schedule which combined "bolus plus infusional" 5-FU compared to "bolus" 5-FU. These results suggest that 24-or 48-hour infusion of high-dose 5-FU is more effective than the conventional bolus schedules.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent or metastatic colorectal adenocarcinoma
* Patients are indicated for 5-FU (1st-line after recurrence/metastasis), OR have failed 5-FU ,treatment with other schedules
* At least one bi-dimensionally measurable lesion(s)
* Previous C/T, R/T >= 4 weeks
* KPS > 50%
* Age >= 18 years
* Fasting TG > 70 mg/dL (within 7 days)
* WBC >= 3,000/uL or ANC >= 1,500/uL
* Plt >= 75,000/uL
* Cre<= 1.5 mg/dL
* Proteinuria < 1+
* Normal T-bil
* AST/ ALT <= 3.5-fold of ULN

Exclusion Criteria:

* Concomitant anticancer therapy or radiotherapy
* CNS metastasis
* Pregnant women
* Patients who have second malignancy
* Symptomatic heart disease (significant arrhythmia, CHF or MI within 3 months of entry)
* Active infection exists
* Extensive liver disease or liver cirrhosis
* Patients who refuse Port-A catheter implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-03; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicity | 2000~2005

SECONDARY OUTCOMES:
response | 2000~2005

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Huei Yeh, M.D., Ph.D., Principal Investigator — Department of Oncology, National Taiwan University hospital
Locations (1):
- Department of Oncology, National Taiwan University hospital, Taipei, Taiwan